CLINICAL TRIAL: NCT02343250
Title: A Randomized, Open-label, Single Dosing, Two-way Crossover Clinical Trial to Compare the Safety/Tolerability and Pharmacokinetics of the Combination of Cilnidipine 10mg and Valsartan 160mg in Comparison to Each Component Coadministered in Healthy Male Volunteers
Brief Title: A Bioequivalence Study Comparing Cilnidipine/Valsartan Combination With Coadministration of Cilnidipine and Valsartan
Acronym: IDCV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-IDCV-103
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — cilnidipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinidipine/Valsartan tablet (Experimental): Cinidipine/Valsartan tablet
  Interventions: Drug: Cilnidipine/Valsartan; Drug: Cilnidipine+Valsartan
- Cilnidipine+Valsartan (Active Comparator): coadministration of cilinidipine and valsartan
  Interventions: Drug: Cilnidipine+Valsartan; Drug: Cilnidipine/Valsartan

INTERVENTIONS:
Drug: Cilnidipine/Valsartan — Cilnidipine 10mg/Valsartan 160mg oral on day1 of 14day cycle
  Arms: Cinidipine/Valsartan tablet
Drug: Cilnidipine+Valsartan — Cinidipine 10mg+Valsartan 160mg oral on day1 of 14day cycle
  Arms: Cilnidipine+Valsartan
Drug: Cilnidipine/Valsartan — Cilnidipine 10mg/Valsartan 160mg oral on day1 of 14day cycle
  Arms: Cilnidipine+Valsartan
Drug: Cilnidipine+Valsartan — Cinidipine 10mg+Valsartan 160mg oral on day1 of 14day cycle
  Arms: Cinidipine/Valsartan tablet

SUMMARY:
A Randomized, Open-label, Single Dosing, Two-way Crossover Clinical Trial to Compare the Safety/Tolerability and Pharmacokinetics of the Combination of Cilnidipine 10mg and Valsartan 160mg in Comparison to Each Component Coadministered in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypertension of hypotension

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
AUClast | 0~24hr
Cmax | 0~24hr

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsang Yu, PhD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- See also: Related Info — http://www.ildong.com